CLINICAL TRIAL: NCT01078129
Title: Efficacy of Hierarchized Computer-assisted Cognitive Remediation Therapy in Schizophrenia
Brief Title: Cognitive Remediation Therapy and Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Collaborators: University Hospital, Grenoble (Other); University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2005-094B
Record Dates: First submitted 2010-02-22; First posted 2010-03-02 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Schizophrenia
Keywords: cognitive deficits
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- behavior therapy - CRT (Active Comparator): behavior program consisting of 14 training sessions of 4 cognitive functions (attention/concentration, topological memory, logical reasoning, executive functions) by means REHACOM® software
  Interventions: Behavioral: cognitive remediation therapy
- non-CRT (Sham Comparator): no intervention
  Interventions: Behavioral: non-CRT

INTERVENTIONS:
Behavioral: cognitive remediation therapy — program consisting of 14 training sessions of 4 cognitive functions (attention/concentration, topological memory, logical reasoning, executive functions)by means REHACOM® software
  Other Names: CRT; behavioral intervention
  Arms: behavior therapy - CRT
Behavioral: non-CRT — waiting list
  Other Names: no intervention
  Arms: non-CRT

SUMMARY:
Objectives:

The purpose of this study is to determine the impact of a new Cognitive Remediation Therapy (CRT) on cognition, social autonomy, symptoms and brain functioning in patients with schizophrenia.

DETAILED DESCRIPTION:
Methods:

In a 2 arms blind study versus sham,80 patients with schizophrenia were enrolled in a program consisting of 14 training sessions of 4 cognitive functions (attention/concentration, topological memory, logical reasoning, executive functions)by means REHACOM® software. Measures of cognitive functioning using the Cogtest® battery as well as social autonomy (Social Autonomy Scale, EAS) and schizophrenia symptoms (Positive And Negative Syndrome Scale, PANSS) were undertaken at the beginning and the end of the meetings of remediation.

Among those 80 participants, 30 patients to (15 active / 15 sham) were randomized to participate in an fMRI study in order to investigate the impact of such CRT program on brain functioning (n-back task before CRT and 3 months later).

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia (DSM IV criteria)
* remitted symptoms
* french language
* informed consent

Exclusion Criteria:

* addiction, neurological disease
* only for second randomized patient participating in MRI study (n=30) : MRI counterindications

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2006-01; Primary Completion 2008-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
cognitive deficits (attention/concentration, topological memory, logical reasoning, executive functions) | before and after CRT (3 months later)
  standardised COGTEST battery (for details see cogtest.com). Cognitive performances were assessed 2 times : at inclusion and 3 months later (after CRT).

SECONDARY OUTCOMES:
brain functioning (fMRI) | before and after CRT (3 months later)
  fMRI during a n-back task, 2 times, before CRT and 3 months later. The 2 sub-groups of 15 patients will be compared with healthy subjects performances at the same task.
schizophrenia symptoms | before CRT and 3 months later
  standardised psychometric scale measuring Positive an Negative Symptoms (PANSS)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry d'amato, MD, PhD, Principal Investigator — Hopital le Vinatier
Locations (1):
- Hôpital le vinatier, Bron, France

REFERENCES:
- [Derived] Bor J, Brunelin J, d'Amato T, Costes N, Suaud-Chagny MF, Saoud M, Poulet E. How can cognitive remediation therapy modulate brain activations in schizophrenia? An fMRI study. Psychiatry Res. 2011 Jun 30;192(3):160-6. doi: 10.1016/j.pscychresns.2010.12.004. Epub 2011 May 2. PMID 21543191